CLINICAL TRIAL: NCT05856812
Title: BOrrelia BUrgdorferi IN Children and Adolescents- a Seroprevalence Study
Brief Title: BOrrelia BUrgdorferi IN Children and Adolescents
Acronym: BOBUINCA
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02143; ks23Heininger
Record Dates: First submitted 2023-04-26; First posted 2023-05-12 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: B. Burgdorferi Infection
Keywords: children; adolescents
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess B. burgdorferi antibodies in children and adolescents in north-western Switzerland and neighbouring countries ("Triregio") treated at the University Children's Hospital Basel to define age-dependent B. burgdorferi seroprevalence rates.

DETAILED DESCRIPTION:
Lyme borreliosis is one of the most prevalent tick-borne zoonosis in the northern hemisphere. Children with Borrelia (B.) burgdorferi infection present with different clinical stages and related symptoms: an early localized stage is commonly associated with an erythema migrans or a borrelial lymphocytoma. Early disseminated disease include early neuroborreliosis, acute arthritis or carditis. Later disease stages include acrodermatitis chronica atrophicans, late neuroborreliosis or Lyme Arthritis. B. burgdorferi prevalence is highest in Europe and has been increasing in the last decade.

Only limited data about the seroprevalence in children is available. A recently published systematic review and meta-analysis estimated the overall global seroprevalence at 14.5% (95% confidence interval (CI) 12.8-16.3%), and at 7.1% (95% CI 5.1-9.5%) in those <40 years of age (based on 18 studies). Only a few studies included in this systematic review assessed paediatric cohorts in Europe: One study from Germany was published 10 years ago and estimated the seroprevalence at 4.5% (95% CI 4.3-5.4%) in the age group 1-17 years. The seroprevalence was higher in males and in the southern part of Germany, and it increased by 11% and 6% for every year of age in boys and girls, respectively. A study from Sweden looked at 5-year old children and estimated a seroprevalence of 3.2%. More data about the seroprevalence is available in adults with heterogenous findings: recent studies from southern Germany, eastern Slovakia, Jordan, Finland and Romania, reported seroprevalence values of 2.4%, 13%, 11.7%, 3.9% and 7.4% respectively.

More recent estimates of the seroprevalence stratified by age are needed in routine care to enable definition of pre-test probability for this serological test in the clinical evaluation of children with suspected Lyme disease. Since an age dependant relationship is plausible and has been shown in studies, seroprevalence estimates from adults should not be used in children. Knowledge of the seroprevalence of B. burgdorferi in children will help to better differentiate between active Lyme disease and seroprevalence due to previous Borrelia infection without signs of active disease. This is also important for avoiding overtreatment of children without active diseases. Only a small amount of plasma or serum is needed to determine the B. burgdorferi antibodies. Therefore, this study aims to evaluate the seroprevalence B. burgdorferi antibodies from left-over blood samples that were taken for other clinically relevant tests without an additional invasive procedure for the child.

ELIGIBILITY:
Inclusion Criteria:

* signed informed general consent
* residence in cantons Basel city, Basel country, Aargau, Solothurn and neighboring areas of France and Germany (Germany postal codes 794x, 795x, 796x, 797x and France postal codes 68480, 68640, 68220, 68330, 68300, 68128, 68730, 68870, 68510, 68130, 68640, 68960, 56890, 68118, 68580, 68680, 68440, 68720)

Exclusion Criteria:

- case blood is taken repetitively from the same child, only the first sample will be used and the child will only be included in the study once.

Refugees seeking asylum will be excluded. These children will be identified by postal address of the Bundesasylzentrum.

* Children presenting for a diagnosis related to a B. burgdorferi infection will be excluded since including these children would result in an over-estimation of the pre-test prevalence of B. burgdorferi IgG due to a possible selection bias. Diagnosis related to a B. burgdorferi infection will include erythema migrans, borrelial lymphocytoma, early or late neuroborreliosis, acute arthritis or carditis, acrodermatitis chronica atrophicans.
* Children with underlying chronic disease, that potentially affects plasma antibodies will be excluded, these include for example the following conditions:

  * known inborn or acquired immunodeficiency syndrome
  * Systemic lupus erythematosus
  * Children with history of intravenous immunoglobulin treatment in the past 12 months for any reason including Kawasaki Disease, Paediatric Inflammatory Multisystem Syndrome, Immunothrombocytopenia.
  * Children after allogenic stem cell transplantation.
  * Children with cancer or known chronic hematology disease.
  * Children treated with immunosuppressive treatment in the last 6 months including systemic steroids >2 weeks duration (>2mg/kg or >20 mg prednisone equivalent) or immunosuppressive combination treatments (e.g. biological disease modifying antirheumatic drugs (DMARDs) + conventional DMARDs), Rituximab or leflunomide

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include children and adolescents, who presented at the University Childrens Hospital Basel in outpatient or inpatient setting.
  All children and adolescents, from whom a sufficient left over amount of the EDTA sample taken for clinical routine tests at the hematology laboratory of the University Childrens Hospital Basel will be included
Sampling Method: Probability Sample
Enrollment: 962 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Assesment of B.burgdorferi antibodies in children and adolescents | one time assessment at baseline
  Analysis of blood samples using B. burgdorferi Immunoglobulin G ELISA test and line blot for confirmation.
  A positive serology for B. burgdorferi will be defined as a positive Immunglobulin G (IgG) enzyme-linked immunoassay (ELISA) test for B. burgdorferi and a positive confirmation test by Line Blot (similar to a western blot technique).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Heininger, Prof., Principal Investigator — University Childrens Hospital
Locations (1):
- University Childrens Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Heeb L, Fritschi N, Marten A, Welzel T, Ritz N, Heininger U. Borrelia burgdorferi infections in children and adolescents in Switzerland - a seroprevalence study 2023/2024 (BOBUINCA). Infection. 2025 Jun;53(3):893-903. doi: 10.1007/s15010-024-02387-7. Epub 2024 Sep 26. PMID 39325354